CLINICAL TRIAL: NCT06192472
Title: Investigation Into the Pathophysiology and Treatment of Varicose Veins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: The Whiteley Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 112453
Record Dates: First submitted 2014-05-20; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins | interventions — Sodium Tetradecyl Sulfate; Polidocanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1% Sodium Tetradecyl Sulphate (Experimental): Superficial leg veins will be removed by phlebectomy operations. Sections of vein 3-5cm in length will be filled with sclerosant.
  Interventions: Procedure: Chemical sclerotherapy; Drug: 1% Sodium Tetradecyl Sulphate
- 3% Sodium Tetradecyl Sulphate (Experimental): Superficial leg veins will be removed by phlebectomy operations. Sections of vein 3-5cm in length will be filled with sclerosant.
  Interventions: Procedure: Chemical sclerotherapy; Drug: 3% Sodium Tetradecyl Sulphate
- 0.5% Polidocanol (Experimental): Superficial leg veins will be removed by phlebectomy operations. Sections of vein 3-5cm in length will be filled with sclerosant.
  Interventions: Procedure: Chemical sclerotherapy; Drug: 0.5% Polidocanol
- 3% Polidcanol (Experimental): Superficial leg veins will be removed by phlebectomy operations. Sections of vein 3-5cm in length will be filled with sclerosant.
  Interventions: Procedure: Chemical sclerotherapy; Drug: 3% Polidcanol

INTERVENTIONS:
Procedure: Chemical sclerotherapy — Sclerosant will be retained within the vein
Drug: 1% Sodium Tetradecyl Sulphate — 1% Sodium Tetradecyl Sulphate
  Arms: 1% Sodium Tetradecyl Sulphate
Drug: 3% Sodium Tetradecyl Sulphate — 3% Sodium Tetradecyl Sulphate
  Arms: 3% Sodium Tetradecyl Sulphate
Drug: 0.5% Polidocanol — 0.5% Polidocanol
  Arms: 0.5% Polidocanol
Drug: 3% Polidcanol — 3% Polidcanol
  Arms: 3% Polidcanol

SUMMARY:
Chemical sclerotherapy is commonly used to treat varicose veins which affect superficial veins in the leg. Sclerotherapy is injected directly into veins where it causes damage to the vein wall. If sufficient damage occurs, the vein is transformed into a fibrous cord which does not re-open. This study will investigate the structural changes caused to the wall of veins following injection with sclerotherapy ex vivo. Vein samples will be obtained from the Whiteley Clinic in Guildford from patients undergoing phlebectomy operations. These will then be injected with sclerotherapy and the extent of damage will be investigated. Samples will also be used for laboratory analysis into the pathophysiology of varicose veins.

DETAILED DESCRIPTION:
Varicose veins affect up to 40% of the population and are associated with significant discomfort, skin damage, and complications including ulceration and perforation. In recent years, there has been a move towards minimally invasive treatment, including chemical sclerotherapy. Despite their widespread use,the fundamental effects of sclerosants have not been fully characterised. Furthermore, their use is associated with significant rates of re-canalisation and clinical recurrence. There is therefore significant scope for researching the effects of sclerosants on the vein wall and the mechanisms of cell death. Furthermore, the pathophysiology of varicose veins has not been fully characterised. It is the aim of this study to research a number of themes related to the use of sclerotherapy and the pathophysiology of varicose veins in order to provide information which will both further scientific knowledge and further develop clinical practice by optimising the use of sclerotherapy. This research will be conducted by a PhD student based at the University of Surrey, in conjunction with the Whiteley Clinic in Guildford. Veins and blood samples removed following varicose vein surgery at the Whiteley Clinic will be provided for laboratory-based research at the university. A range of methodologies will be employed to analyse cellular responses to sclerosants to determine the precise structural and biochemical changes which lead to destruction of the vein and clinical efficacy, and to investigate a number of key themes implicated in the pathophysiology of varicose veins.

ELIGIBILITY:
Inclusion Criteria:

* Gives consent
* Over 18 years
* Undergoing phlebectomy operation

Exclusion Criteria:

* Does not give consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
To identify the mechanisms responsible for the therapeutic effects of sclerotherapy in varicose veins. | 2 years 4 months
  no additional details - project ended 2015 and staff have left

SECONDARY OUTCOMES:
To gain further insight into the pathological mechanisms underlying varicose vein formation and recurrence, and to identify a biomarker which indicates susceptibility to development of varicose veins. | 2 years 4 months
  no additional details - project ended 2015 and staff have left

CONTACTS AND LOCATIONS:
Overall Officials: Christopher T Lee, MPharm, Principal Investigator — Univesity of Surrey; Jian-Mei Li, MBBS MD PhD, Study Director — University of Surrey; Mark S Whiteley, MS, Study Director — The Whiteley Clinic and University of Surrey
Locations (2):
- United Kingdom (2):
  - The Whiteley Clinic, Guildford, Surrey
  - University of Surrey, Guildford, Surrey